CLINICAL TRIAL: NCT05544734
Title: Analysis of Hydrocodone Compared to Acetaminophen and Ibuprofen for Post-nail Procedure Analgesia
Brief Title: Hydrocodone Compared to Acetaminophen and Ibuprofen for Post-nail Procedure Analgesia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21-10024054
Record Dates: First submitted 2022-09-13; First posted 2022-09-16 (Actual); Results first posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Nail Diseases; Nail Abnormality
Keywords: nail diseases; nail biopsy; nail procedure; pain management
MeSH Terms: conditions — Nail Diseases; Nails, Malformed; Agnosia | interventions — Hydrocodone; Acetaminophen; acetaminophen, hydrocodone drug combination; oxycodone-acetaminophen; Ibuprofen

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Hydrocodone 5mg/acetaminophen 325mg (Active Comparator): Participants receive oral hydrocodone 5 mg/acetaminophen 325 mg every 4 hours for 2 days, followed by oral acetaminophen 1000 mg and oral ibuprofen 400 mg every 6 hours for 4 days
  Interventions: Drug: Hydrocodone 5Mg/Acetaminophen 325Mg Tab; Drug: Acetaminophen 1000mg; Drug: Ibuprofen 400 mg
- Acetaminophen 1000mg + Ibuprofen 400mg (Active Comparator): Participants receive oral acetaminophen 1000 mg and oral ibuprofen 400 mg every 6 hours for 6 days
  Interventions: Drug: Acetaminophen 1000mg; Drug: Ibuprofen 400 mg

INTERVENTIONS:
Drug: Hydrocodone 5Mg/Acetaminophen 325Mg Tab — 5 mg/325 mg tablet
  Other Names: Vicodin; Norco; Lortab
  Arms: Hydrocodone 5mg/acetaminophen 325mg
Drug: Acetaminophen 1000mg — 1000 mg tablet
  Other Names: Tylenol
Drug: Ibuprofen 400 mg — 400 mg tablet
  Other Names: Advil; Motrin

SUMMARY:
The purpose of this study is to assess the safety and efficacy of ropivacaine and hydrocodone for nail-procedure associated pain management. The investigators hypothesize that ropivacaine with hydrocodone will be superior to ropivacaine with acetaminophen and ibuprofen for managing pain.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing fingernail or toenail, excision, or shave biopsy
* Must understand and voluntarily sign an informed consent form
* Must be male or female and aged 18-95 years at time of consent
* Must be able to adhere to the study visit schedule and other protocol requirements

Exclusion Criteria:

* Subject is unable to provide written informed consent for any reason
* Subject has peripheral vascular disease, arterial insufficiency, peripheral neuropathy
* Subject is on Aspirin, NSAIDs, or consumes a chronic medication for control of any other chronic pain
* Subject has a history of opioid or alcohol use disorder
* Subject has a history of peptic ulcer disease, gastritis, chronic renal insufficiency or a history of kidney disease, or has underlying liver disease
* Subject has a history of severe constipation
* Subject is sensitive or allergic to any of the elements included in this study
* Subject is unable to complete the required pain dairy
* Subject is pregnant, planning pregnancy, or nursing

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-11-10 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2023-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shari Lipner, MD, PhD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Medical College of Cornell University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hwang JK, Ricardo JW, Lipner SR. Combination of acetaminophen and ibuprofen is noninferior to acetaminophen and hydrocodone for postnail procedure analgesia: A randomized controlled trial. J Am Acad Dermatol. 2023 Dec;89(6):1300-1302. doi: 10.1016/j.jaad.2023.08.042. Epub 2023 Aug 22. No abstract available. PMID 37619705

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Hydrocodone 5mg/Acetaminophen 325mg | Acetaminophen 1000mg + Ibuprofen 400mg
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hydrocodone 5mg/Acetaminophen 325mg | Acetaminophen 1000mg + Ibuprofen 400mg | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 7 | 13
  >=65 years | 4 | 3 | 7
Age, Continuous [Mean (Full Range); unit: years] | 53.3 [22 to 84] | 47.7 [23 to 69] | 50.5 [22 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 4 | 4 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 6
  Not Hispanic or Latino | 7 | 7 | 14
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 7 | 6 | 13
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Pain Scores on Postoperative Day 2, as Measured by the Wong-Baker 0-to-10 Pain Scale
Description: Change in pain scores obtained with the Wong-Baker 0-to-10 pain scale between the 2 groups on postoperative day 2. The Wong-Baker 0-to-10 pain scale is used for rating the severity of pain, with scores ranging from 0 to 10, and higher scores indicating greater severity of pain.
Time Frame: Baseline, 2 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Hydrocodone 5mg/Acetaminophen 325mg | Acetaminophen 1000mg + Ibuprofen 400mg
Number analyzed (Participants) | 10 | 10
score on a scale | 2.1 (1.6) | 2.4 (1.7)
Statistical Analysis 1: Comparison: Hydrocodone 5mg/Acetaminophen 325mg vs Acetaminophen 1000mg + Ibuprofen 400mg; Test type: Superiority; p = 0.69, t-test, 2 sided; Median Difference (Final Values) = -0.30, 95% CI 2-sided [-1.85 to 1.25] — Direction = Hydrocodone group mean change (i.e., change = baseline to postoperative day 2) minus Non-Hydrocodone group mean change (i.e., change = baseline to postoperative day 2)

2. Secondary Outcome: Change in Health-related Quality of Life Scores on Postoperative Days 3 and 6, as Measured by an Adapted APS-POQ-R Questionnaire
Description: Change in health-related quality of life associated with pain obtained with an adapted version of the APS-POQ-R (APS Patient Outcome Questionnaire) between the 2 groups on postoperative days 3 and 6. The APS-POQ-R is a questionnaire used for rating health-related quality of life associated with pain, with scores of each domain ranging from 0 to 10 or 0% to 100%, and higher scores indicating greater severity of impact on quality of life (12 domains summed up for total score range of minimum 0 to maximum 120).
Time Frame: 3 days, 6 days (end of study)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Hydrocodone 5mg/Acetaminophen 325mg | Acetaminophen 1000mg + Ibuprofen 400mg
Number analyzed (Participants) | 10 | 10
score on a scale | 12.7 (11.2) | 10.4 (9.0)
Statistical Analysis 1: Comparison: Hydrocodone 5mg/Acetaminophen 325mg vs Acetaminophen 1000mg + Ibuprofen 400mg; Test type: Superiority; p = 0.62, t-test, 2 sided; Median Difference (Final Values) = 2.30, 95% CI 2-sided [-7.25 to 11.85] — Direction = Hydrocodone group mean change (i.e., change = postoperative day 3 to postoperative day 6) minus Non-Hydrocodone group mean change (i.e., change = postoperative day 3 to postoperative day 6)

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Hydrocodone 5mg/Acetaminophen 325mg | Acetaminophen 1000mg + Ibuprofen 400mg
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-15): https://cdn.clinicaltrials.gov/large-docs/34/NCT05544734/Prot_SAP_000.pdf